CLINICAL TRIAL: NCT01956409
Title: Use of Proton MR Spectroscopy and 18F-Fluorocholine PET for Breast Cancer Diagnosis, Prediction of Clinical Outcome and Monitoring of Treatment Response to Neoadjuvant Chemotherapy
Brief Title: Proton MR Spectroscopy and 18F-Fluorocholine PET for Breast Cancer Diagnosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201201056MIB
Record Dates: First submitted 2013-09-25; First posted 2013-10-08 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer Diagnosis; Positron Emission Tomography; Magnetic Resonance Imaging
Keywords: breast neoplasms; 18F-FCH PET; MRI
MeSH Terms: conditions — Breast Neoplasms | interventions — fluorocholine; Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diagnostic accuracy of PET and MR spectroscopy (Experimental): To investigate the diagnostic accuracy of 18F-Fluorocholine PET and proton MR spectroscopy of breast lesions, using pathology as gold standard.
  Interventions: Drug: 18F-FCH; Drug: Magnevist

INTERVENTIONS:
Drug: 18F-FCH
  Other Names: N,N-Dimethyl-N-Fluoromethylethanolamine
Drug: Magnevist
  Other Names: Gadopentetate dimeglumine

SUMMARY:
The application of FCH PET in breast cancer diagnosis has not been reported.

We hypothesize that FCH reveals choline metabolic profiles of breast cancers, and shows the similar pathophysiological mechanism to choline on proton MRS, and our study goals are:

1. To investigate and compare the diagnostic performance of proton MRS and FCH PET for localized findings on mammography and breast ultrasound.
2. To investigate whether FCH PET findings are correlated with choline signals on proton MRS.
3. To evaluate if choline, water and lipid signals on proton MRS, FCH PET are associated with factors related to clinical outcome and prognosis- that is, molecular markers, tumor staging, histologic grade of breast cancers.
4. For localized advanced breast cancer, to investigate the treatment response to NAC using proton MRS and FCH PET, and to evaluate which modality is more sensitive.
5. To investigate the usefulness of FCH PET for whole body staging for breast cancer patients.

DETAILED DESCRIPTION:
In recent years, the application of 18F-FDG PET (positron emission tomography) and MRI for breast lesion diagnosis was emerging. Imbriaco et al compared the diagnostic performance of 18F-FDG PET and MRI for suspicious breast lesions, with PET showing a sensitivity of 80% and specificity 100%; and MRI revealed a sensitivity of 95% and specificity of 98%. Lim et al studied 18F-FDG PET-CT with MRI to monitor treatment response for breast cancer patients receiving NAC, with a sensitivity 70% and specificity 72%, and can detect the treatment response earlier than conventional imaging.

However, 18F-FDG is not tumor specific, and searching for an alternative tracer agent as a tumor biomarker is necessary. 18F-Fluorocholine (FCH), a choline analog, was used for diagnosis of prostate cancer, hepatocellular carcinoma (HCC), bronchioloalveolar carcinoma, brain tumor, since malignant tumors show higher choline metabolites than benign lesions; it was reported that FCH PET showed higher sensitivity (88-94%) than 18F-FDG PET (59-68%) in detecting HCC. FCH PET was used for staging for prostate cancer, with FCH PET-CT can provide sufficient information for management with an accuracy of 88%.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-75 years old.
* with localized findings on mammography or breast ultrasound in recent 3 months and who will receive breast biopsy or excision for the findings; or with recently diagnosed LABC who will receive NAC.

Exclusion Criteria:

* unable to cooperate with the examinations
* pregnant or planning to be pregnant
* estimated GFR (eGFR) < 60 ml/min/1.73m2 or with recent acute renal failure, past history of renal dialysis.
* Past history of claustrophobia
* Past history of anaphylactoid reactions to MRI contrast agents or PET tracer agents.
* with cardiac pacemaker, aneurysmal clip, mechanical valve replacement, recently applied coronary artery stent (<2 months).
* Past history of breast cancer or other malignancy (treated within 5 years).
* lactating.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of 18F-FCH PET for breast cancer diagnosis | 5 years
  The investigators use the interpretation results of 18F-FCH PET for breast lesion diagnosis, with the pathology result of the breast lesions as gold standards, and to investigate how well the 18F-FCH PET can correctly diagnose the true nature of breast lesions.

SECONDARY OUTCOMES:
Monitoring of treatment response of breast cancer to chemotherapy using 18F-FCH PET | 5 years
  For the breast cancer patients who will undergo chemotherapy treatment, we aim to use 18F-FCH PET before and after chemotherapy. And the changes of tracer uptake of 18F-FCH on PET scans before and after chemotherapy will be correlated with clinical outcomes before and after chemotherapy, to investigate whether 18F-FCH PET results can monitor treatment response of chemotherapy.
diagnostic accuracy of breast MR spectroscopy for breast cancer diagnosis | 5 years
  The investigators use the interpretation results of breast MRI (with MR spectroscopy in the examination) for breast lesion diagnosis, with the pathology result of the breast lesions as gold standards, and to investigate how well the breast MRI study can correctly diagnose the true nature of breast lesions.

OTHER OUTCOMES:
Evaluation the correlation of 18F-FCH PET and breast MRI | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jane Wang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan